CLINICAL TRIAL: NCT05645978
Title: Association of Obesity and Cardiovascular Outcomes in Patients With Pacemaker : a Korean Nationwide Cohort Study
Brief Title: Association of Obesity and Cardiovascular Outcomes in Patients With Pacemaker
Acronym: Paradox
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ajou University School of Medicine (Other)
Responsible Party: Principal Investigator, Kwang-No Lee, Professor, Ajou University School of Medicine
Other Study IDs: AJOUIRB-EXP-2021-398-6
Record Dates: First submitted 2022-12-02; First posted 2022-12-12 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Pacemaker Complication; Arrhythmias, Cardiac; Obesity; Cardiovascular Morbidity
Keywords: Pacemaker; Obesity paradox
MeSH Terms: conditions — Arrhythmias, Cardiac; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients who underwent pacemaker insertion during study period: Patients who underwent pacemaker insertion between January 2015 and December 2020
  Interventions: Device: Pacemaker insertion

INTERVENTIONS:
Device: Pacemaker insertion — Patients who underwent pacemaker insertion between January 2015 and December 2020
  Other Names: Insertion of pacemaker

SUMMARY:
In this study, the investigators evaluated the association between various measures of adiposity [BMI and waist circumference (WC)] and clinical outcomes in Asian patients who underwent pacemaker insertion, using a nationwide population based cohort.

DETAILED DESCRIPTION:
This retrospective nationwide cohort study used administrative claims data from the Korean National Health Insurance Service (NHIS) and the combined health check-up database of the National Health Insurance Corporation between 2013 and 2020.

The investigators included patients who underwent pacemaker insertion between January 2015 and December 2020. Patients aged <20 years, those who were already taken pacemaker insertion before 2015, and those with cancer were excluded from the analysis. The follow-up period was defined as the time from the index date (date of device procedure) to each outcome event, date of death, or end of the study period (December 31, 2020), whichever came first.

Patients' demographic data, comorbidities, concomitant medications, and income level were collected from the Korean NHIS database. The recent health check-up data from the index date was also ascertained, including height, weight, waist circumference, blood pressure, health surveys, and laboratory exam. Health survey included family history, smoking history, alcohol history, and the level of individual physical activity.

According to BMI following the World Health Organization recommendation for Asian population, study patients were categorized into 5 groups: underweight, <18.5 kg/m2; normal range, 18.5 to <23 kg/m2; overweight, 23 to <25 kg/m2; obese I, 25 to <30 kg/m2; and obese II, ≥30 kg/m2[4]. The investigators defined the proportion of medical use by calculating formula with the recuperation cost and the number of the visit to hospitals.

During the follow-up period, the investigators assessed 3 clinical outcomes, including all-cause death, cardiovascular hospitalization and the recurrence rate. Clinical outcomes were mainly defined by the the International Classification of Diseases, 10th revision (ICD-10). Patients were censored at the clinical outcomes or the end of the study period (December 31, 2020), whichever came first.

All categorical variables are presented as frequencies and percentages. Normally distributed data were presented as mean ± standard deviation, whereas nonparametric data are presented as median and interquartile range by BMI.

Cox proportional hazard regression analyses were performed to identify the association of BMI with the primary and secondary outcomes, calculating hazard ratio (HR) and 95% confidence interval (CI) and adjusting for the following potential confounders: sex, age, systolic blood pressure, fasting glucose level, total cholesterol level, alcohol consumption, smoking status, physical activity, household income, use of antihypertensive agents, use of statins, use of antiplatelet agents, previous history of MI, previous history of stroke, and index year. All analyses were conducted using R-statistics.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent pacemaker insertion between January 2015 and December 2020

Exclusion Criteria:

* Patients aged <20 years
* Patients already taken pacemaker insertion before 2015
* Patients with cancer

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We included patients who underwent pacemaker insertion between January 2015 and December 2020. Patients aged <20 years, those who were already taken pacemaker insertion before 2015, and those with cancer were excluded from the analysis. The follow-up period was defined as the time from the index date (date of device procedure) to each outcome event, date of death, or end of the study period (December 31, 2020), whichever came first.
Sampling Method: Non-Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Composite of Outcomes | 5 years
  Death + CV hospitalization + Fatal arrest event + Infective endocarditis

SECONDARY OUTCOMES:
Death | 5 years
  Mortality
CV hospitalization | 5 years
  Admission caused by Cardiovacular disease
Fatal arrest event | 5 years
  Event of cardiac arrest by ventricular tachycardia and fibrillation
Infective endocarditis | 5 years
  Diagnosed with infective endocarditis

CONTACTS AND LOCATIONS:
Overall Officials: Kwang-No LEE, Study Chair — Ajou University School of Medicine
Locations (1):
- Ajou University School of Medicine, Suwon, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kim MS, Kim WJ, Khera AV, Kim JY, Yon DK, Lee SW, Shin JI, Won HH. Association between adiposity and cardiovascular outcomes: an umbrella review and meta-analysis of observational and Mendelian randomization studies. Eur Heart J. 2021 Sep 7;42(34):3388-3403. doi: 10.1093/eurheartj/ehab454. PMID 34333589
- [Background] Prasitlumkum N, Chokesuwattanaskul R, Kaewput W, Thongprayoon C, Bathini T, Boonpheng B, Vallabhajosyula S, Cheungpasitporn W, Jongnarangsin K. Utilization and in-hospital complications of catheter ablation for atrial fibrillation in patients with obesity and morbid obesity. Clin Cardiol. 2022 Apr;45(4):407-416. doi: 10.1002/clc.23795. Epub 2022 Feb 16. PMID 35170775
- [Background] Seo J, Li W, Safiriyu I, Kharawala A, Nagraj S, Tahir A, Doundoulakis I, Koliastasis L, Rios S, Palaiodimos L, Kokkinidis DG. A Meta-Analysis on the Impact of High BMI in Patients Undergoing Transcatheter Aortic Valve Replacement. J Cardiovasc Dev Dis. 2022 Nov 9;9(11):386. doi: 10.3390/jcdd9110386. PMID 36354785